CLINICAL TRIAL: NCT06895031
Title: A Multi-center, Open-label, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of JYP0015 in Advanced Solid Tumors With RAS Mutation
Brief Title: Study of JYP0015 in Patients With Advanced Solid Tumors Harboring Specific Mutations in RAS
Acronym: STAR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JYP0015M101
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor; Pancreatic Ductal Adenocarcinoma (PDAC); Non-small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC)
Keywords: PDAC; NSCLC; CRC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JYP0015 in RAS-Mutant Solid Tumors (Experimental): This arm includes participants with histologically or pathologically confirmed advanced solid tumors harboring RAS mutations, identified via molecular testing. RAS mutations are defined as nonsynonymous mutations in KRAS, NRAS, or HRAS at codons 12, 13, 61, 117, or 146 (e.g., G12, G13, Q61, K117, or A146). Participants will receive JYP0015 as an oral tablet.
  Interventions: Drug: JYP0015

INTERVENTIONS:
Drug: JYP0015 — JYP0015 is an orally bioavailable pan-RAS inhibitor designed to target the active (ON) form of wild-type and mutant RAS across KRAS, NRAS, and HRAS isoforms. The drug will be administered orally, with dosing determined by the study protocol in the dose-escalation and indication-expansion phases.

SUMMARY:
Evaluate the safety and antitumor activity of JYP0015 in adults with specific RAS mutant advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1/2, multicenter, open-label study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and clinical activity of JYP0015 in adult patients with advanced solid tumors harboring specific RAS mutations.

The study consists of two parts:

* Phase 1 (dose escalation) - Evaluates the safety, tolerability, and pharmacokinetic profile of JYP0015 monotherapy, preliminarily assesses efficacy, and determines the recommended dose (RD) for further evaluation.
* Phase 2 (indication expansion) - Explores the therapeutic potential of JYP0015 monotherapy at the RD across four predefined cohorts:

  1. Pancreatic ductal adenocarcinoma (PDAC)
  2. Non-small cell lung cancer (NSCLC)
  3. Colorectal cancer (CRC)
  4. Other advanced solid tumors Phase 2 will assess both efficacy and safety within these cohorts.

JYP0015 is a potent, orally bioavailable pan-RAS inhibitor that selectively targets the active (ON) form of wild-type and mutant RAS across all three isoforms-HRAS, NRAS, and KRAS.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or pathologically confirmed solid tumors with RAS mutation via molecular tests.
2. Patients with RAS mutation who have disease progression or intolerance after adequate standard treatment
3. Eastern Cooperative Oncology Group (ECOG) performance status in 0 or 1
4. Adequate organ function

Exclusion Criteria:

1. Presence of central nervous system (CNS) metastases; however, subjects with previously treated brain metastases may be enrolled if clinically stable.
2. Gastrointestinal (GI) disorders that may interfere with drug administration/absorption, including but not limited to: Dysphagia or inability to swallow tablets， Malabsorption syndrome，Refractory nausea, vomiting, or diarrhea，Chronic GI diseases (e.g., Crohn's disease, ulcerative colitis)
3. Congestive heart failure with New York Heart Association (NYHA) functional class ≥II or left ventricular ejection fraction (LVEF) <50%.
4. Any other condition deemed by the investigator to potentially compromise study outcomes or lead to premature termination, including but not limited to: Alcohol or substance abuse，Concurrent severe medical conditions (e.g., psychiatric disorders requiring active treatment)， Familial or social circumstances that may affect patient safety, compliance, or study data collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicity (DLT) | 21 days
  The number of participants experiencing dose-limiting toxicities (DLT) during the dose-escalation period of the study.
Incidence and Severity of Treatment-Emergent Adverse Events (AEs) and Serious AEs | Up to 3 years
  The incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including abnormalities in laboratory values and vital signs.
Overall Response Rate (ORR) | Up to 3 years
  Overall response rate assessed per RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Maximum Observed Blood Concentration (Cmax) of JYP0015 | Up to 16 weeks
  Maximum plasma concentration (Cmax) of JYP0015 following administration.
Time to Reach Maximum Blood Concentration (Tmax) of JYP0015 | Up to 16 weeks
  Time to reach maximum plasma concentration (Tmax) of JYP0015 following administration.
Duration of Response (DOR) | Up to 3 years
  Duration of response as assessed by RECIST v1.1.
Time to Response (TTR) | Up to 3 years
  Time to response as assessed by RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No